CLINICAL TRIAL: NCT02492542
Title: Effect of Pelvic Floor Stimulation on the Pelvic Floor Function in Cervical Cancer Patients With Type III Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wang Jianliu (Other)
Collaborators: Peking University (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Beijing Hospital (Other Government); Chinese PLA General Hospital (Other); Peking University Cancer Hospital & Institute (Other); Chinese Academy of Medical Sciences (Other); Beijing Obstetrics and Gynecology Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor-Investigator, Wang Jianliu, Peking University People's Hospital Ob and Gy, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D151100001915003
Record Dates: First submitted 2015-06-25; First posted 2015-07-08 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: electrical stimulation; urinary incontinence
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electric Stimulation Treatment (Experimental): Patients in the intervention group were treated with electric stimulation based on the routine clinical nursing.
  Interventions: Device: PHENIX USB 8.
- control group (No Intervention): patients in this group only received routine clinical nursing without electric stimulation

INTERVENTIONS:
Device: PHENIX USB 8. — Electrical stimulation program: frequency: 1/4/Hertz (HZ), pulse width: 270/230/270 μs, time: 30min. Electrode piece: 50*50mm sticky electrode plate. Position: an electrode piece is placed in the S3, and an electrode piece is placed in the bladder region.Current intensity adjusted according to the patient's tolerance, the maximum current intensity of the pain was not appropriate, generally not more than 100milliampere(mA).Devices PHENIX USB 8.
  Other Names: Electric Stimulation Treatment
  Arms: Electric Stimulation Treatment

SUMMARY:
The purpose of this study is to investigate the effect of electric stimulation on the pelvic floor function in cervical cancer patients with type III hysterectomy.

DETAILED DESCRIPTION:
This is a prospective, multi center, open, randomized, controlled clinical trial. All cervical carcinoma patients who undergo type III hysterectomy in the hospitals involved in this study were recruited. 5-7 days postoperative, those who meet the inclusion criteria and without the exclusion criteria and sign the consent were randomized grouped of intervention and control objective by 1:1. At the same time, according to the research hospital, menopausal status (menopause vs menopause) and surgery approach (laparoscopic vs open)，they were further stratified randomly. Patients in the intervention group received electrical stimulation treatment based on conventional clinical nursing, while patients in control group only receive routine clinical care. Except for the treatment of electrical stimulation, other research procedures is the same in the two groups. The recovery rate of urination function, pelvic floor function and life quality of the two group is compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as cervical squamous cell carcinoma on Ⅰa2, Ib1 or Ⅱa1 stage
* Type III hysterectomy
* There are pathological results showing that cancer resection clean and no distant metastasis,Specifically as follows:Lymph nodes(-);cancer foci invasion depth <1/2;Lymphatic space(-);Vaginal stump(-);differentiation G1-2.
* Patients agreed to the study, informed consent

Exclusion Criteria:

* Radiotherapy and chemotherapy before surgery
* Reserved nerve in the surgery
* Urinary system damage
* POP(Pelvic Organ Prolapse stage)>II stage before surgery
* Moderate above stress urinary incontinence(SUI) before surgery(1 hours urine pad test>=10g)
* Urinary retention before surgery
* Severe constipation or difficult defecation before surgery
* There are uncontrolled epilepsy, central nervous system disease or mental disorder history in patients.The clinical severity of these diseases Influence clinical research compliance,judging by the researcher.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Urination function recovery rate | From 14 days to 24 months after operation

SECONDARY OUTCOMES:
Number of participants with recovery of defecation function and urinary function after III hysterectomy | From 14 days to 24 months after operation
Quality of life Questionnaire | From 14 days to 24 months after operation
Overall Survival | From 14 days to 24 months after operation
  The overall survival (OS) in cervical cancer patients after 3 years' III hysterectomy after comparison of pelvic floor rehabilitation therapy and control group
Disease-free survival | From 14 days to 24 months after operation
  Comparison of pelvic floor rehabilitation treatment group and control group of cervical cancer patients with type III hysterectomy 3 years disease-free survival (DFS)

CONTACTS AND LOCATIONS:
Overall Officials: Wang J liu, Doctor, Study Chair — Peking University People's Hospital Ob and Gy

REFERENCES:
- [Result] Plotti F, Angioli R, Zullo MA, Sansone M, Altavilla T, Antonelli E, Montera R, Damiani P, Benedetti Panici P. Update on urodynamic bladder dysfunctions after radical hysterectomy for cervical cancer. Crit Rev Oncol Hematol. 2011 Nov;80(2):323-9. doi: 10.1016/j.critrevonc.2010.12.004. Epub 2011 Jan 31. PMID 21277788
- [Result] Griffenberg L, Morris M, Atkinson N, Levenback C. The effect of dietary fiber on bowel function following radical hysterectomy: a randomized trial. Gynecol Oncol. 1997 Sep;66(3):417-24. doi: 10.1006/gyno.1997.4797. PMID 9299255
- [Result] Raspagliesi F, Ditto A, Fontanelli R, Zanaboni F, Solima E, Spatti G, Hanozet F, Vecchione F, Rossi G, Kusamura S. Type II versus Type III nerve-sparing radical hysterectomy: comparison of lower urinary tract dysfunctions. Gynecol Oncol. 2006 Aug;102(2):256-62. doi: 10.1016/j.ygyno.2005.12.014. Epub 2006 Jan 30. PMID 16445968
- [Result] Jackson KS, Naik R. Pelvic floor dysfunction and radical hysterectomy. Int J Gynecol Cancer. 2006 Jan-Feb;16(1):354-63. doi: 10.1111/j.1525-1438.2006.00347.x. PMID 16445658
- [Result] Sood AK, Nygaard I, Shahin MS, Sorosky JI, Lutgendorf SK, Rao SS. Anorectal dysfunction after surgical treatment for cervical cancer. J Am Coll Surg. 2002 Oct;195(4):513-9. doi: 10.1016/s1072-7515(02)01311-x. PMID 12375757
- [Result] Axelsen SM, Petersen LK. Urogynaecological dysfunction after radical hysterectomy. Eur J Surg Oncol. 2006 May;32(4):445-9. doi: 10.1016/j.ejso.2006.01.017. Epub 2006 Mar 3. PMID 16516431
- [Result] Butler-Manuel SA, Summerville K, Ford A, Blake P, Riley AJ, Sultan AH, Monga AK, Stanton SL, Shepherd JH, Barton DP. Self-assessment of morbidity following radical hysterectomy for cervical cancer. J Obstet Gynaecol. 1999 Mar;19(2):180-3. doi: 10.1080/01443619965552. PMID 15512265
- [Result] Manchana T, Sirisabya N, Lertkhachonsuk R, Worasethsin P, Khemapech N, Sittisomwong T, Vasuratna A, Termrungruanglert W, Tresukosol D. Long term complications after radical hysterectomy with pelvic lymphadenectomy. J Med Assoc Thai. 2009 Apr;92(4):451-6. PMID 19374292
- [Result] Sansone M, Plotti F, Panici PB. Long-term lower urinary tract dysfunction after radical hysterectomy in patients with early postoperative voiding dysfunction. Int Urogynecol J. 2010 Oct;21(10):1309-10; author reply 1311-2. doi: 10.1007/s00192-010-1206-1. Epub 2010 Jun 23. No abstract available. PMID 20571765
- [Result] Barnes W, Waggoner S, Delgado G, Maher K, Potkul R, Barter J, Benjamin S. Manometric characterization of rectal dysfunction following radical hysterectomy. Gynecol Oncol. 1991 Aug;42(2):116-9. doi: 10.1016/0090-8258(91)90329-4. PMID 1894168
- [Result] Ye S, Yang J, Cao D, Lang J, Shen K. A systematic review of quality of life and sexual function of patients with cervical cancer after treatment. Int J Gynecol Cancer. 2014 Sep;24(7):1146-57. doi: 10.1097/IGC.0000000000000207. PMID 25033255
- [Result] Maddocks M, Lewis M, Chauhan A, Manderson C, Hocknell J, Wilcock A. Randomized controlled pilot study of neuromuscular electrical stimulation of the quadriceps in patients with non-small cell lung cancer. J Pain Symptom Manage. 2009 Dec;38(6):950-6. doi: 10.1016/j.jpainsymman.2009.05.011. PMID 19748761
- [Result] Bennett MI, Johnson MI, Brown SR, Radford H, Brown JM, Searle RD. Feasibility study of Transcutaneous Electrical Nerve Stimulation (TENS) for cancer bone pain. J Pain. 2010 Apr;11(4):351-9. doi: 10.1016/j.jpain.2009.08.002. Epub 2009 Oct 22. PMID 19853518
- [Result] Robb K, Oxberry SG, Bennett MI, Johnson MI, Simpson KH, Searle RD. A cochrane systematic review of transcutaneous electrical nerve stimulation for cancer pain. J Pain Symptom Manage. 2009 Apr;37(4):746-53. doi: 10.1016/j.jpainsymman.2008.03.022. Epub 2008 Sep 14. PMID 18790600
- [Result] Yang EJ, Lim JY, Rah UW, Kim YB. Effect of a pelvic floor muscle training program on gynecologic cancer survivors with pelvic floor dysfunction: a randomized controlled trial. Gynecol Oncol. 2012 Jun;125(3):705-11. doi: 10.1016/j.ygyno.2012.03.045. Epub 2012 Apr 1. PMID 22472463
- [Result] Ryu JS, Kang JY, Park JY, Nam SY, Choi SH, Roh JL, Kim SY, Choi KH. The effect of electrical stimulation therapy on dysphagia following treatment for head and neck cancer. Oral Oncol. 2009 Aug;45(8):665-8. doi: 10.1016/j.oraloncology.2008.10.005. Epub 2008 Dec 17. PMID 19095492
- [Derived] Wang S, Gao L, Wen H, Gao Y, Lv Q, Li H, Wang S, Wang Y, Liu Q, Han J, Wang H, Li Y, Yu N, Wang Q, Cao T, Wang S, Sun H, Wang Z, Sun X, Wang J. Evaluation of pelvic floor muscle function (PFMF) in cervical cancer patients with Querleu-Morrow type C hysterectomy: a multicenter study. Arch Gynecol Obstet. 2022 Feb;305(2):397-406. doi: 10.1007/s00404-021-06290-6. Epub 2021 Oct 28. PMID 34713337
- [Derived] Li XW, Gao L, Wang Q, Lv QB, Xia ZJ, Wen HW, Han JS, Wu YM, Wang SM, Liu Q, Li H, Wang HB, Li Y, Wang SY, Wang ZQ, Sun XL, Wang JL. Long-Term Effect of Early Post-operative Transcutaneous Electrical Stimulation on Voiding Function After Radical Hysterectomy: A Multicenter, Randomized, Controlled Trial. Front Med (Lausanne). 2021 Sep 30;8:677029. doi: 10.3389/fmed.2021.677029. eCollection 2021. PMID 34660617
- [Derived] Sun XL, Wang HB, Wang ZQ, Cao TT, Yang X, Han JS, Wu YF, Reilly KH, Wang JL. Effect of transcutaneous electrical stimulation treatment on lower urinary tract symptoms after class III radical hysterectomy in cervical cancer patients: study protocol for a multicentre, randomized controlled trial. BMC Cancer. 2017 Jun 15;17(1):416. doi: 10.1186/s12885-017-3387-1. PMID 28619043